CLINICAL TRIAL: NCT04490395
Title: Increasing Physical Resilience in Older Adults With Osteoarthritis Pain: Feasibility and Acceptability of a Brief Behavioral Physical Activity Intervention
Brief Title: Increasing Physical Activity in Older Adults With Osteoarthritis Pain: Examining a Brief Behavioral Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105573
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Engage PA; treatment as usual
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engage PA (Experimental)
  Interventions: Behavioral: Engage PA
- Treatment as usual plus fitness tracker (Other)
  Interventions: Other: Treatment as Usual plus (TAU+)

INTERVENTIONS:
Behavioral: Engage PA — Engage PA will consist of a 2-session intervention delivered to participants at the medical center or virtual visit by their study therapist, and includes a wearable personal fitness monitor for tracking their daily activity levels throughout.
  Arms: Engage PA
Other: Treatment as Usual plus (TAU+) — The comparison condition will receive treatment as usual throughout the study, and are given a wearable personal fitness monitor for tracking their daily activity levels throughout the study.
  Arms: Treatment as usual plus fitness tracker

SUMMARY:
The purpose of this study is to evaluate how older adults might benefit from sessions that teach behavioral coping skills for increasing physical activity and reducing interference from arthritis pain. This study will randomize individuals to receive Engage-PA, or continue to receive treatment as usual. Engage-PA involves two sessions (about 45 minutes each) with a study therapist that teaches individuals behavioral skills for increasing daily steps. These behavioral skills include identifying their personal values and instructions on how to pace their daily physical activity to avoid creating severe pain when walking. All participants in the study will wear small devices that track physical activity such as daily steps throughout the study, which also allow participants to see their daily step counts and overall level of activity. All participants will answer a set of questions about how much arthritis gets the way of many important life activities, their success at living in line with their personal values, and how much thoughts, feelings and body sensations get in the way of living a satisfying life. These questions will be asked at the beginning of the study and 6 weeks into the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* English speaking
* Diagnosis of osteoarthritis in knee or hip
* Able to ambulate even if assisted with ambulatory device such as walker or cane
* Endorse worst pain and pain interference as ≥ 3 out of 10 within the last week

Exclusion Criteria:

* Planned surgery during study duration that would limit mobility (e.g., due to recommended rehabilitation or recovery period) for more than 3 weeks
* Current enrollment in cardiac rehabilitation
* Myocardial infarction in the past 3 months
* Major surgery requiring limited movement or mobility for recovery within the past 3 months
* Presence of a serious psychiatric condition (e.g., schizophrenia, suicidal intent) indicated by medical chart, treating medical provider or other staff, or study staff interactions that would contraindicate safe study participation
* Medical provider indicating that exercise (even walking) should only be medically supervised; as determined by medical record review or patient reported
* Fall or falls within the last 3 months that led to immediate medical treatment/hospitalization
* Reported or suspected moderate or severe cognitive impairment subsequently informed by a Folstein Mini-Mental Status Examination of <19

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Plumb Vilardaga, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plumb Vilardaga JC, Kelleher SA, Diachina A, Riley J, Somers TJ. Linking physical activity to personal values: feasibility and acceptability randomized pilot of a behavioral intervention for older adults with osteoarthritis pain. Pilot Feasibility Stud. 2022 Aug 1;8(1):164. doi: 10.1186/s40814-022-01121-0. PMID 35915512
- [Derived] Vilardaga JCP, Kelleher S, Diachina A, Riley J, Somers T. Linking Physical Activity to Personal Values: Feasibility and Acceptability Randomized Pilot of a Behavioral Intervention for Older Adults with Osteoarthritis Pain. Res Sq [Preprint]. 2022 Jan 3:rs.3.rs-1182374. doi: 10.21203/rs.3.rs-1182374/v1. PMID 35018370

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Started | 19 | 20
Completed | 19 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.32 (6.01) | 71.20 (4.42) | 71.55 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 12 | 12 | 24
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled in the Study
Description: How many participants, up to the expected 40 participants, enroll in the study within the study period
Time Frame: 9 months
Population: Expected participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 20 | 20
Participants | 19 | 20

2. Primary Outcome: Number of Participants Who Completed the Entire Program
Description: Participants who complete all assessments and required study sessions
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 19 | 20
Participants | 19 | 20

3. Primary Outcome: Percentage of Participants Who Were Mostly or Very Satisfied With the Intervention
Description: Client Satisfaction Questionnaire asks 12 questions related to patient satisfaction on a Likert scale of 1 = very satisfied to 7 = very dissatisfied. There is one item assessing overall satisfaction with the intervention, and the percentage of participants responding to this item with "mostly" or "very" satisfied is reported below.
Time Frame: Post treatment (6 weeks)
Population: Only those receiving the active treatment (Engage PA group) were given this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Engage PA
Number analyzed (Participants) | 18
percentage of participants | 89

4. Secondary Outcome: Arthritis Pain (AIMS 2 Symptom Subscale)
Description: The Arthritis Impact Measurement Scale (AIMS 2) measures arthritis pain related disability across areas of living both with a total score and on several subscales (i.e., pain severity, physical functioning/pain-related disability, psychological distress), where 1 indicates very good functioning, and 5 indicates very poor functioning. Symptom subscale includes items assessing pain severity, stiffness, and physical discomfort. Range is 5 to 25 where higher scores indicate worse functioning.
Time Frame: Baseline, post-treatment (6 weeks)
Population: Data not collected (n=1; TAU group) due to lost to follow up, data not analyzed (n=1; Engage PA group) due to assessment conducted out of window.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 13.72 (3.80) | 14.90 (4.16)
  Post-Treatment | 11.78 (3.69) | 14.58 (4.50)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority; p = 0.044, t-test, 2 sided; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [-0.26 to 3.62]

5. Secondary Outcome: Arthritis-related Physical Functioning (AIMS 2 Physical Functioning Subscale)
Description: The Arthritis Impact Measurement Scale (AIMS 2) measures arthritis pain related disability across areas of living on several subscales (i.e., pain severity, physical functioning/pain-related disability, psychological distress), where 1 indicates very good functioning, and 5 indicates very poor functioning. Physical functioning subscale includes items assessing mobility level, walking and bending, self-care and household tasks. Range is 5-25 where higher scores indicate worse functioning.
Time Frame: Baseline, post-treatment (6 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 6.38 (1.89) | 7.44 (2.00)
  Post-Treatment | 6.64 (1.38) | 7.51 (2.09)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority; p = 0.056, t-test, 2 sided; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-0.15 to 1.33]

6. Secondary Outcome: Psychological Distress (AIMS 2 Affect Subscale)
Description: The Arthritis Impact Measurement Scale (AIMS 2) measures arthritis pain related disability across areas of living on several subscales (i.e., pain severity, physical functioning/pain-related disability, psychological distress), where 1 indicates very good functioning, and 5 indicates very poor functioning. Psychological distress subscale includes items assessing mood and anxiety/tension. Range is 5-25 where higher scores indicate worse functioning.
Time Frame: Baseline, post-treatment (6 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 10.36 (3.12) | 10.37 (2.85)
  Post-treatment | 10.59 (4.15) | 10.33 (2.18)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority; p = 0.377, t-test, 2 sided; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.75 to 1.28]

7. Secondary Outcome: Daily Step Count in 7 Day Period
Description: Daily step counts as reported to study staff, after participants recorded them from wearable fitness trackers at end of day. Each assessment period consisted of 7 continuous days of wear. Summed totals of steps in the 7 day period were calculated, and then means calculated between groups of these summed step counts for the 7 day assessment period.
Time Frame: Baseline, post-treatment (6 weeks)
Population: Only some participants were able to record daily steps data due to complications with devices and COVID-19 protocols.
Measure: Mean (Standard Deviation); unit: Mean of total steps in 7 day period
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 9 | 9
Mean of total steps in 7 day period
  Baseline | 35712.55 (27441.78) | 28165.89 (20916.05)
  Post-treatment | 38268.56 (28154.68) | 28154.67 (29183.00)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Only 9 cases had any data available per group, and some had missing values and were not included in each analysis; Test type: Superiority — Within subjects change over time; p = 0.258, ANOVA; Change over time; F test (1,15) df = 1.381; Within subjects change over time
Statistical Analysis 2: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority — Between group analysis; p = 0.627, ANOVA; F test (1,15) df = 0.246; Between group analysis
Statistical Analysis 3: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Time x Condition interaction; Test type: Superiority; p = 0.947, ANOVA; F test (1,15) df = 0.005; Time x Condition interaction

8. Secondary Outcome: Rapid Assessment of Physical Activity
Description: The RAPA is a self-reported measure that assesses participants engagement in a variety of activities, such as light movement, moderate activity, vigorous activity, and other activities such as strength-training or yoga. Scores range from 0 - 7, where higher scores indicate greater involvement in physical activity overall.
Time Frame: Baseline, post-treatment (6 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 3.25 (1.22) | 3.16 (1.50)
  Post-treatment | 3.47 (1.73) | 2.31 (1.19)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority; p = 0.038, t-test, 2 sided; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.85 to 0.98]

9. Secondary Outcome: Psychological Flexibility
Description: The Acceptance and Action Questionnaire-II asks about psychological flexibility, defined as how often thoughts, feelings and body sensations get in the way of living a fulfilling life. Responses are on a 1 to 7 Likert scale with 1 indicating that these issues never get in the way, and 7 indicating that these issues always get in the way. Range is 7 - 49, with lower scores indicating better outcomes.
Time Frame: Baseline, post-treatment (6 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 13.95 (8.20) | 16.21 (7.45)
  Post-Treatment | 14.72 (8.37) | 13.05 (6.31)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority; p = 0.07, t-test, 2 sided; Mean Difference (Final Values) = -2.56, 95% CI 2-sided [-6.05 to 0.94]

10. Secondary Outcome: Valued Living - Health Domain
Description: The Bulls-Eye Values measure assesses how successfully participants are at living in line with 4 domains of personal values (relationships, leisure, health, and work) on a visual dart-board scale with 1 indicating perfect success, and 14 indicates being unsuccessful. Range for each domain is 1 - 14 with lower as better outcome.
Time Frame: Baseline, post-treatment (6 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 4.11 (2.26) | 4.05 (1.99)
  Post-treatment | 3.76 (1.44) | 4.88 (1.73)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority; p = 0.43, t-test, 2 sided; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-1.19 to 1.42]

11. Secondary Outcome: Valued Living - Leisure Domain
Description: as for outcome 10
Time Frame: Baseline, post-treatment (6 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 4.26 (2.26) | 4.60 (4.18)
  Post-treatment | 4.12 (1.87) | 4.18 (2.01)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority; p = 0.72, t-test, 2 sided; Mean Difference (Final Values) = -.029, 95% CI 2-sided [-.194 to 1.42]

12. Secondary Outcome: Valued Living - Relationship Domain
Description: The Bulls-Eye Values measure assesses how successfully participants are at living in line with 4 domains of personal values (relationships, leisure, health, and work) on a visual dart-board scale with 1 indicating perfect success, and 14 indicates being unsuccessful.
Time Frame: Baseline, post-treatment (6 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 3.68 (2.11) | 4.29 (2.29)
  Post-treatment | 4.00 (2.10) | 4.35 (2.15)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority; p = 0.341, t-test, 2 sided; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.35 to 0.23]

13. Secondary Outcome: Valued-Living - Work/Community Domain
Description: as for outcome 12
Time Frame: Baseline, post-treatment (6 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 3.32 (1.97) | 3.30 (1.87)
  Post-Treatment | 3.65 (2.03) | 3.41 (2.24)
Statistical Analysis 1: Comparison: Engage PA vs Treatment as Usual Plus Fitness Tracker; Test type: Superiority; p = 0.25, t-test, 2 sided; Mean Difference (Final Values) = -.059, 95% CI 2-sided [-2.35 to 1.17]

ADVERSE EVENTS:
Time Frame: Approximately 6 weeks
Arm/Group | Engage PA | Treatment as Usual Plus Fitness Tracker
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

LIMITATIONS AND CAVEATS:
Changes to measurement type during trial due to pandemic-related challenges (no objective daily steps data available despite intention to collect this data).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT04490395/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT04490395/ICF_000.pdf